CLINICAL TRIAL: NCT03719534
Title: An Open-label, Multicenter, Randomized, Phase 3 Trial to Assess the Efficacy and Safety of Coinfusion With Unrelated Cord Blood Unit for Patients With Acute Myeloid Leukemia Undergoing Haploidentical Hematopoietic Cell Transplantation
Brief Title: Haplo HCT vs Haplo-cord HCT for Patients With AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Zhejiang University (Other); The Second People's Hospital of Huai'an (Other); Soochow Hopes Hematology Hospital (Unknown); Hygeia Suzhou Yongding Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ3703
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hematopoietic Stem Cell Transplantation; Haplo-identical Donor; Cord Blood Unit; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-HCT (Active Comparator): people enrolled in this arm will receive a typical haploidentical donor HCT
  Interventions: Procedure: haplo-HCT
- Haplo-cord HCT (Experimental): people enrolled in this arm will receive a coinfusion of cord blood unit in addition to a typical haploidentical donor HCT
  Interventions: Procedure: haplo-cord HCT

INTERVENTIONS:
Procedure: haplo-HCT — HCT will be performed with a haploidentical donor
  Arms: Haplo-HCT
Procedure: haplo-cord HCT — Haploidentical donor HCT will be performed with coinfusion of unrelated cord blood unit
  Arms: Haplo-cord HCT

SUMMARY:
Patients who have acute myeloid leukemia and will undergo haplo-identical donor hematopoeitic cell transplantation (haplo HCT) are potential candidates of this trial. Participants will randomized into two arms: Arm A will undergo a typical haplo HCT, while Arm B will receive an coinfusion of an unrelated cord blood unit (haplo-cord HCT) in addition to Arm A. Progression-free survival, overall survival, cumulative incidence of relapse and nonrelapse mortality will be recorded as endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years old;
2. Patients with AML;
3. With available minimal residual disease (MRD) parameters assessed by flow cytometry (FCM) and/or quantitative real-time PCR (qPCR)
4. Having no available HLA-matched donor, and willing to undergo haplo-HCT and having a suitable haploidentical donor
5. With Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
6. Signing informed consent form, having the ability to comply with study and follow-up procedures

Exclusion Criteria:

1. Acute promyelocytic leukaemia (AML subtype M3)
2. With other malignances
3. Failing to acquire a suitable UCB unit
4. With previous history of autologous haematopoietic cell transplantation (auto-HCT), allogeneic haematopoietic cell transplantation (allo-HCT) or chimaeric antigen receptor T-cell therapy
5. With uncontrolled infection intolerant to haplo-HCT
6. With severe organ dysfunction

   * Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
   * Respiratory failure (PaO2≤60 mmHg)
   * Hepatic abnormalities (total bilirubin≥2×upper limit of normal [ULN], alanine aminotransferase or aspartate aminotransferase≥2×ULN)
   * Renal dysfunction (creatinine≥2 mg/dL creatinine clearance rate < 30 mL/min)
7. In pregnancy or lactation period
8. With any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 year after randomization
  estimated overall survival at 3 year

SECONDARY OUTCOMES:
Progression-free survival | 3 year after randomization
  estimated progression-free survival at 3 year
Cumulative incidence of relapse | 3 year after randomization
  estimated cumulative incidence of nonrelapse mortality at 3 year
Cumulative incidence of non-relapse mortality | 3 year after randomization
  estimated nonrelapse mortality at 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (5):
- China (5):
  - The Second People's Hospital of Huai'an, Huai'an, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Soochow Hopes Hematology Hospital, Suzhou, Jiangsu
  - Hygeia Suzhou Yongding Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou B, Chen J, Liu T, Ye Y, Zhang Y, Ding Y, Liu H, Zhu M, Ma X, Li X, Zhao L, Lin Z, Huang H, Xu Y, Wu D. Haploidentical hematopoietic cell transplantation with or without an unrelated cord blood unit for adult acute myeloid leukemia: a multicenter, randomized, open-label, phase 3 trial. Signal Transduct Target Ther. 2024 May 6;9(1):108. doi: 10.1038/s41392-024-01820-5. PMID 38705885